CLINICAL TRIAL: NCT07124624
Title: Impact of an AI-Driven CT Angiography Model on Intracranial Aneurysm Detection and Clinical Outcomes in Regional Hospitals (IDEAL2): A Nationwide Stepped-Wedge Cluster-Randomized Trial
Brief Title: Stepped-Wedge Cluster Randomized Trial of AI-Assisted CTA Detection for Intracranial Aneurysms in Regional Hospitals
Acronym: IDEAL2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang longjiang,MD, Head of Radiology, Jinling Hospital, China
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025DZKY-087-01
Record Dates: First submitted 2025-08-07; First posted 2025-08-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Aneurysm; CT Angiography; AI (Artificial Intelligence); Cluster Randomized Trial
Keywords: Intracranial aneurysm; AI (Artificial Intelligence); Stepped-wedge cluster-randomized trial
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Assisted Diagnosis (Experimental): Patients in this group will undergo head CTA, interpreted by radiologists with the assistance of a previously validated deep learning AI model. The model highlights suspected aneurysm candidates on the CTA images to support diagnostic decision-making.
  Interventions: Device: AI-Assisted CTA Interpretation
- Standard Diagnosis (Active Comparator): Patients in this group will undergo head CTA, which will be interpreted by radiologists following standard local diagnostic protocols. No AI assistance will be provided during image interpretation.
  Interventions: Diagnostic Test: Standard CTA Interpretation

INTERVENTIONS:
Device: AI-Assisted CTA Interpretation — A locked, independently validated deep learning model was used to assist radiologists in interpreting head CTA scans. The model was trained on 16,546 CTA cases and externally validated on an independent set of 900 DSA-verified CTA cases, achieving a patient-level sensitivity of 0.943 and an average of 0.187 false positives per case.
  Arms: AI-Assisted Diagnosis
Diagnostic Test: Standard CTA Interpretation — Head CTA interpretation performed by radiologists using local routine diagnostic workflows without AI support.
  Arms: Standard Diagnosis

SUMMARY:
This study (IDEAL 2) is a nationwide stepped-wedge cluster-randomized trial designed to prospectively enroll over 14,400 patients undergoing outpatient head CT angiography (CTA). The trial will be conducted across more than 72 regional hospitals in China. Clusters were randomly assigned to nine randomization groups. In accordance with the stepped-wedge design, clusters will sequentially transition from the control condition (standard human diagnosis) to the intervention condition (AI-assisted diagnosis) at regular intervals over a 10-month period, until all clusters receive the intervention. The primary outcome is the detection rate of intracranial aneurysms. Secondary outcomes include patient prognosis and clinical outcomes.

DETAILED DESCRIPTION:
A multicenter, stepped-wedge cluster-randomized trial will be conducted in regional hospitals, specifically prefecture-level and county-level institutions across China. Each cluster (i.e., hospital) will enroll approximately 200 patients undergoing head computed tomography angiography (CTA), yielding a total sample size of at least 14,400 participants. The trial consists of nine steps, each lasting one month. Clusters will transition sequentially from the control condition to the intervention condition based on stratified randomization, until all clusters have received the intervention.

In the control group, diagnoses and treatments will follow local standard clinical protocols. In the intervention group, diagnostic procedures will be supported by an artificial intelligence (AI)-assisted system. The primary outcome is the detection rate of intracranial aneurysms, as determined from radiology reports at the patient level. Secondary outcomes include additional diagnostic performance metrics on CTA, such as the detection of intracranial arterial stenosis, occlusion, and tumors.

Follow-up evaluations at 3 and 12 months will assess treatment-related indicators-including repeat head CTA or magnetic resonance angiography (MRA), hospitalization rates, and digital subtraction angiography (DSA) utilization-as well as clinical outcomes related to aneurysm events. These measures aim to evaluate both the short- and long-term impacts of AI-assisted diagnosis on routine clinical practice and patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

-Patients in the outpatient setting who are scheduled to undergo head CTA scanning

Exclusion Criteria:

* Age < 18 years
* History of cerebrovascular surgery involving any metallic implants (e.g., aneurysm embolization, aneurysm clipping, or vascular stenting)
* Modified Rankin Scale (mRS) score > 3
* Refuse to sign written informed consent
* Contraindications to CTA examination
* CTA scan failure, incomplete imaging data, or image quality insufficient for diagnostic evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14400 (Estimated)
Dates: Start 2025-10-09 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of intracranial aneurysms | Day 1
  The proportion of patients diagnosed with intracranial aneurysms among all individuals undergoing CTA during the observation period. This outcome is used to compare the diagnostic effectiveness of conventional radiologist interpretation based on local clinical practice versus AI-assisted diagnosis in detecting intracranial aneurysms.

SECONDARY OUTCOMES:
Detection rates of other intracranial lesions except aneurysms | Day 1
  The proportion of patients diagnosed with intracranial arterial stenosis, occlusion, arteriovenous malformation (AVM), Moyamoya disease, or other vascular abnormalities among all individuals undergoing CTA during the observation period.
Follow-up visits and referrals | At 3-month and 12-month follow-up.
  The number of follow-up or referral visits, including the number of follow-up visits, number of referrals, and repeated noninvasive vascular imaging examinations (e.g., CTA, MRA, or high-resolution vessel wall MRI).
Hospitalization | At 3-month and 12-month follow-up.
  Subsequent hospitalization outcomes during patient follow-up, including the rate of hospitalization, rate of hospitalization specifically related to intracranial aneurysms and the length of hospital stay.
Invasive DSA examinations | At 3-month and 12-month follow-up.
  Rate of patients undergoing digital subtraction angiography (DSA), along with the distribution of findings, including positive identification of aneurysms, other vascular abnormalities, or no detectable abnormalities.
Aneurysm treatment decisions | At 3-month and 12-month follow-up.
  Distribution of aneurysm management strategies, including conservative treatment, endovascular coiling, surgical clipping, and other approaches.
Intraoperative complications | At 3-month and 12-month follow-up.
  The rate of aneurysm treatment-related complications-such as intraoperative rupture, , vasospasm, neurological injury, and other adverse events.
Postoperative complications | At 3-month and 12-month follow-up.
  Postoperative complications, including cerebral edema, intracranial hematoma, hydrocephalus, and recurrent thrombosis.
In-hospital morbidity | At 3-month and 12-month follow-up.
  In-hospital morbidity, defined as a Modified Rankin Scale (mRS) score of 3-5 at hospital discharge. The Modified Rankin Scale ranges from 0 to 6, with higher scores indicating greater disability (scores of 3-5) or death (score of 6).
In-hospital mortality | At 3-month and 12-month follow-up.
  In-hospital mortality, defined as a Modified Rankin Scale (mRS) score of 6 at hospital discharge. The Modified Rankin Scale ranges from 0 to 6, with a score of 6 indicating death.
All-cause mortality | At 3-month and 12-month follow-up.
  All-cause mortality during patient follow-up.
Aneurysm-related events during follow-up | At 12-month follow-up.
  Proportion of patients with aneurysm-related events during follow-up, including aneurysm growth (≥1 mm in any dimension), aneurysm rupture (non-traumatic subarachnoid hemorrhage), stroke (hemorrhagic or ischemic), de novo aneurysm formation, and aneurysm recurrence after treatment.

IPD SHARING:
Plan to Share IPD: No